CLINICAL TRIAL: NCT02210793
Title: Evaluation of Dry Eye Following Transepithelial Photorefractive Keratectomy in Comparison to Conventional LASIK: a Comparative Study
Brief Title: Dry Eye Evaluation After Transepithelial PRK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AL-Nour Eye Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Sherif, Dr Ahmed Sherif, AL-Nour Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ANH-1; ANH-TPRK1 (Other: Al-Nour Eye hospital)
Record Dates: First submitted 2014-08-02; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Dry Eye
Keywords: Transepithelial PRK; Dry eye; Schirmer test; Tear break up time; Dry eye after advanced surface ablation technique
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transepithelial PRK (Active Comparator): 20 eyes to undergo a no touch , all-laser advanced surface ablation technique termed transepithelial PRK using the Amaris laser platform (Schwind eye-tech solutions Gmbh, Germany)
  Interventions: Procedure: transepithelial PRK
- Conventional LASIK (Active Comparator): 20 eyes to undergo LASIK using a mechanical microkeratome (M2, Moria Surgical, Antony, France) and the Mel 80 excimer laser system(Carl Zeiss Meditec)
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: transepithelial PRK
  Arms: Transepithelial PRK
Procedure: LASIK
  Arms: Conventional LASIK

SUMMARY:
The aim of the study is to evaluate the severity of dry eye syndrome following excimer laser vision correction using no-touch all-laser photorefractive keratectomy in comparison to conventional lasik

DETAILED DESCRIPTION:
Prospective interventional clinical study 2 groups: Group A : 20 eyes of 10 patients undergoing transepithelial PRK Group B: 20 eyes of 10 patients undergoing LASIK using mechanical microkeratome Tear Break Up Time and Schirmer 2 tests are used to evaluate severity of dry eye before surgery and 1 , 3 and 6 months postoperative Follow up period : 6 months

ELIGIBILITY:
Inclusion Criteria

* Myopia -1 to -6 diopters
* Astigmatism -0.5 to - 4 diopters

Exclusion Criteria:

* Pregnancy and lactation
* Keratoconus
* Previous refractive surgery
* Previous herpetic keratitis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
qualitative assessment of dry eye syndrome | 6 months
  Tear Break Up time is used as a qualitative measure of dry eye after surgery
quantitative of dry eye after surgery | 6 months
  Schirmer test is used as a quantitative measure of dry eye after surgery

SECONDARY OUTCOMES:
haze | 6 months
  haze is a known possible complication of surface ablation Its severity can be graded according to a slit lamp scoring system

OTHER OUTCOMES:
healing time of epithelial defect epithelial defect | 2-5 days
  the period of time in days needed for complete healing of the epithelial defect created during transepithelial PRK

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shalaby, MD, Study Director — Cairo University; Mahmoud H Abu Steit, MD, Study Director — Cairo University; Mohamed Salah, MBBCH, Study Director — Cairo University
Locations (1):
- Al Nour Eye Hospital, Giza, Egypt